CLINICAL TRIAL: NCT03996681
Title: A Prospective Clinical Trial of TACE Combined With Methylcantharidimide Tablets in the Treatment of Large and Unresectable Hepatocellular Carcinoma
Brief Title: TACE Combined With Methylcantharidimide Tablets in the Treatment of Large and Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suzhou Municipal Hospital (Other)
Responsible Party: Principal Investigator, Lei Chen, vice president of hospital, Suzhou Municipal Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190124R0
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Transarterial Chemoembolization; Methylcantharidimide; Large and unresectable HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — cantharidin methylimide

STUDY DESIGN:
Intervention Model Description: TACE plus methylcantharidimide tablets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE plus methylcantharidimide tablets (Experimental): Methylcantharidimide tablets( 75mg po tid) is administered before first TACE 3 days and taken continuously after TACE treatment. Every 6 weeks is a cycle.
  Interventions: Drug: methylcantharidimide tablets

INTERVENTIONS:
Drug: methylcantharidimide tablets — Drug: methylcantharidimide tablets
  Methylcantharidimide is a single molecule drug used for the treatment of primary liver cancer.
  Procedure: TACE
  Transcatheter arterial chemoembolization was performed by the injection of small embolic particles coated with chemotherapeutic agents selectively into an artery directly supplying a tumor.
  Other Names: GANYU

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of transarterial chemoembolization (TACE) combined with methylcantharidimide tablets in the treatment of patients with large and unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
Most guidelines recommend transarterial chemoembolization (TACE), as the standard of care for unresectable hepatocellular carcinoma (HCC ) at Barcelona Clinic Liver Cancer (BCLC) stage A-B. While a number of studies demonstrate poor effect of TACE for patients with large hepatocellular carcinoma. The efficacy of TACE on large (≥ 10 cm) stage A-B HCC is far from satisfactory. The median overall survival was only 6.5-9.1 months. Methylcantharidimide is a single molecule drug used for the treatment of primary liver cancer.

Thus, the investigators carried out this prospective trial to demonstrate the efficacy and safety of TACE combined with methylcantharidimide tablets in patients with large and unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18-75 years;
2. KPS≥70;
3. The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL);
4. Simultaneously staged as BCLC A or BCLC B based on Barcelona Clinic Liver Cancer staging system;
5. Patients must have at least one tumor lesion that can be accurately measured;
6. Solitary tumor with diameter ≥10cm, or multiple tumors, diameter of the largest was more than 7cm;
7. Diagnosed as unresectable with consensus by the panel of liver surgery experts,
8. Re commanded treated by TACE with consensus by the panel of liver multi-disciplinary treatment (MDT);
9. No past history of TACE, chemotherapy or molecule-targeted treatment;
10. No Cirrhosis or cirrhotic status of Child-Pugh class A only;
11. No liver protection therapy in 2 weeks before enrolled, and meet the following laboratory parameters:(a) Platelet count ≥ 75,000/μL; (b)Hemoglobin ≥ 8.5 g/dL;(c) Total bilirubin ≤ 30mmol/L;(d) Serum albumin ≥ 32 g/L;(e) Glutamic pyruvic transaminase (ALT) and glutamic oxalacetic transaminase (AST) ≤ 6 x upper limit of normal;(f) Serum creatinine≤ 1.5 x upper limit of normal;(g) international normalized ratio（INR）> 2.3 or prothrombin time (PT)/activated partial thromboplastin time (APTT) within normal limits; (h) Absolute neutrophil count (ANC) >1,500/mm3;
12. Ability to understand the protocol and to agree to sign a written informed consent document.

Exclusion Criteria:

1. Factors that affect oral administration, such as dysphagia, chronic diarrhea and intestinal obstruction;
2. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry;
3. Known of serious heart disease which can nor endure the treatment such as cardiac ventricular arrhythmias requiring anti-arrhythmic therapy;
4. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy;
5. Known history of HIV;
6. History of organ allograft;
7. Known or suspected allergy to the investigational agents or any agent given in association with this trial;
8. Evidence of bleeding diathesis;
9. Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug;
10. Serious non-healing wound, ulcer, or bone fracture;
11. Known central nervous system tumors including metastatic brain disease;
12. Poor compliance that can not comply with the course of treatment and follow up;
13. Factors that the researchers consider it not appropriate to be included

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-07-20 (Estimated); Primary Completion 2020-07-20 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 18 months
  DCR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR), or stable disease (SD). CR was defined as disappearance of any intratumoral arterial enhancement in all target lesions. PR was defined as at least a 30% decrease in the sum of diameters of viable (enhancement of arterial phase) target lesions taking as reference the baseline sum of the diameters of target lesions. SD was when a case does not qualify for either PR or progressive disease (PD) and was new non-target lesions. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions.

SECONDARY OUTCOMES:
Time to progression (TTP) | 18 months
  TTP was defined as the time from the date of treatment to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST). Disease progression was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the baseline sum of diameters of target lesions.
Overall Survival (OS) | 18 months
  From the date of treatment until the date of death from any cause
Health Related Quality of Life (HRQoL) | 18 months
  HRQoL assessed using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) .The EORTC QLQ-C30 included 30 questions comprising 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social) and 9 symptom scales (fatigue, pain, nausea/vomiting, dyspnoea, appetite loss, insomnia, constipation, diarrhea and financial difficulties) and a single global health and quality of life status score. Most questions used a 4-point scale (1=Not at all to 4=Very much); 2 questions used a 7-point scale (1= Very poor to 7=Excellent). All domain scores were calculated as an average of item scores and transformed to 0 to 100 score range. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/quality of life (QoL) represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problem.
clinical symptoms | 18 months
  A questionnaire about the clinical symptoms, appetite，pain and sleep.
Adverse Events | 18 months
  Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Lei Chen, MD, Principal Investigator — Suzhou Municipal Hospital
Locations (1):
- Suzhou Municipal Hospital, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in a publication
Time Frame: starting 6 months after publication
Access Criteria: Case Report Form (CRF)

REFERENCES:
- [Background] He MK, Le Y, Li QJ, Yu ZS, Li SH, Wei W, Guo RP, Shi M. Hepatic artery infusion chemotherapy using mFOLFOX versus transarterial chemoembolization for massive unresectable hepatocellular carcinoma: a prospective non-randomized study. Chin J Cancer. 2017 Oct 23;36(1):83. doi: 10.1186/s40880-017-0251-2. PMID 29061175
- [Background] Xue T, Le F, Chen R, Xie X, Zhang L, Ge N, Chen Y, Wang Y, Zhang B, Ye S, Ren Z. Transarterial chemoembolization for huge hepatocellular carcinoma with diameter over ten centimeters: a large cohort study. Med Oncol. 2015 Mar;32(3):64. doi: 10.1007/s12032-015-0504-3. Epub 2015 Feb 15. PMID 25682389
- [Background] Huang YH, Wu JC, Chen SC, Chen CH, Chiang JH, Huo TI, Lee PC, Chang FY, Lee SD. Survival benefit of transcatheter arterial chemoembolization in patients with hepatocellular carcinoma larger than 10 cm in diameter. Aliment Pharmacol Ther. 2006 Jan 1;23(1):129-35. doi: 10.1111/j.1365-2036.2006.02704.x. PMID 16393290
- [Background] Poon RT, Ngan H, Lo CM, Liu CL, Fan ST, Wong J. Transarterial chemoembolization for inoperable hepatocellular carcinoma and postresection intrahepatic recurrence. J Surg Oncol. 2000 Feb;73(2):109-14. doi: 10.1002/(sici)1096-9098(200002)73:23.0.co;2-j. PMID 10694648